CLINICAL TRIAL: NCT02970591
Title: The Role of CARbohydrates in Irritable Bowel Syndrome (CARIBS): Protocol for a Randomized Controlled Trial Comparing Three Different Treatment Options
Brief Title: A Comparison of Three Different Treatment Options for Irritable Bowel Syndrome
Acronym: CARIBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Simrén, Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Car-IBS 1511-01
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: FODMAPS; carbohydrates; metabolomics; microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Diet A (Experimental): Low carbohydrate diet
  Interventions: Other: Traditional dietary advice and low FODMAP content
- Medical treatment (Active Comparator): Optimized Medical treatment
  Interventions: Other: Optimized Medical treatment
- Diet B (Experimental): Traditional dietary advice and low FODMAP content
  Interventions: Other: Low carbohydrate diet

INTERVENTIONS:
Other: Traditional dietary advice and low FODMAP content — Traditional dietary advice according to the Brittish Dietetic Association including reducing the intake of fermentable carbohydrates.
  Arms: Diet A
Other: Low carbohydrate diet — Diet that contains a maximum of 10 energy percent of carbohydrates, 23 energy % proteins and 67 energy % fat.
  Arms: Diet B
Other: Optimized Medical treatment — Standard consultation by physician and if needed patients will receive medical treatment based on the most prominent symptom. Constipation: osmotic laxatives, linaclotide. Diarrhea: loperamid, bile acid binders. Pain: anti depressent, antispasmodics, linaclotide.
  Arms: Medical treatment

SUMMARY:
Irritable Bowel Syndrome is a common disease to which there is no curable treatment. Diet is considered to trigger symptoms associated with the clinical picture of IBS, and dietary treatment is thus believed to relieve the symptoms of IBS. As the disease is very heterogeneous in its manifestation, different treatment options might be indicated depending on the predominant symptom. To investigate the response to different dietary treatment options, a randomized controlled intervention trial will be carried out in adult patients (>18 y) with IBS according to Rome IV criteria. The aim of this study is to compare the response to two different dietary treatments or optimized medical treatment.

DETAILED DESCRIPTION:
The study is a randomized controlled trial comparing three different treatments during four weeks:

1. Combination of low FODMAP diet + traditional dietary advice (based on NICE recommendations)

   * Eat at regular hours; 3 main meals and 3 snacks
   * Eat in peace, chew the food properly
   * Peel all fruits and vegetables
   * Limit intake of spicy and fatty foods, coffe, alcohol, avoid fizzy drinks and chewing gum
   * Choose soluble rather than insoluble fibres
   * Avoid foods high in FODMAPs
2. Diet low in carbohydrates

   * 10 E% carbohydrates, 23 E% protein, 67 E% fat
   * Larger amounts of fish, shellfish, meat, egg, dairy products (lactose free if wanted) nuts, seeds, oil, vegetables
   * No sugary or starchy foods, e.g pasta, potatoes, bread, rice, most fruits
   * No specific consideration about FODMAP content
3. Optimized pharmacological tretament based on predominant symptom and previous experience with pharmacological treatmment.

Pain/discomfort:

* Pain: Amitriptyline 25 mg. Increase to 50 mg if needed
* Episodic pain: Hyoscyamine 0,2mg 2x2; adjust dose if needed
* Pain with diarrhea: Amitriptyline 25 mg. Increase dose if needed
* Pain with constipation: Linaclotide 290 microgram 1x1

Constipation:

* Bulking agent (Sterculia gum (Inolaxol) 1x1. Increase to 1x3 if needed
* Osmotic laxative (Macrogol (Movicol) 1x1
* Linaclotide 290 microgram 1x1 Diarrhea
* Loperamide 1x2 . Adjust dose if needed
* Cholestyramine 1x1. Increase ever 3-5 d as needed
* Ondansetron 4mg 1x1. Increase to 1x2-3 if needed
* Eluxadoline 100mg 1x2

Primary endpoint: IBS-SSS reduction >50 points

ELIGIBILITY:
Inclusion Criteria:

* IBS according to ROME IV criteria, BMI 18-35, ability to communicate in Swedish, Gothenburg region resident

Exclusion Criteria:

* Heart, liver, neurologic or psychiatric disease or illness
* Serious gastrointestinal diseases
* Celiac disease
* Diabetes
* Other conditions or surgery that affects the gastrointestinal function
* Hyperlipidemia
* Food allergy or intolerance other than lactose
* Adherence to a specific diet
* Being pregnant or breastfeeding
* Previously been treated with any of the intervention arms, including having tested all of the pharmacological treatment options of relevance for the symptom profile of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-01; Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
The proportion (%) of patients who respond to treatment | Baseline to 4 weeks
  A responder is defined as having an IBS-SSS reduction >50 points @ 4 weeks

SECONDARY OUTCOMES:
Change in symptom severity | Baseline, 4 weeks, 3 and 6 months
  Absolute and percentage change in IBS-SSS
Determinants for GI symptoms by IBS-SSS | Baseline, 4 weeks, 3 and 6 months
  GI symptoms measured by IBS-SSS
Determinants for GI symptoms by GSRS-IBS | Baseline, 4 weeks, 3 and 6 months
  GI symptoms measured by GSRS-IBS
Predictors of response to treatment | Baseline to 4 weeks
  Potential predictors include demographics, questionnaire data, microbiota, metabolites, immunology
Adherence to allocated intervention | Baseline, 4 weeks, 3 and 6 months
  Including compliance to dietary intervention during 4 weeks, and long-term adherence during follow-up
Change in microbiota content | Baseline, 4 weeks, 6 months
  Fecal microbiota analysis using 16S technique
Change in extra-intestinal symptoms and quality of life | Baseline, 4 weeks, 3 and 6 months
  As assessed by IBS specific questionnaires
Change in metabolic profile | Baseline, 4 weeks, 6 months
  Metabolomics in serum and urine samples

OTHER OUTCOMES:
Qualitative assessment | Approx. at 3 months follow-up
  Patient's subjective experiences related to the dietary intervention described by qualitative methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Magnus Simren, Gothenburg, Non-US/Non-Canadian, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nybacka S, Tornblom H, Josefsson A, Hreinsson JP, Bohn L, Frandemark A, Weznaver C, Storsrud S, Simren M. A low FODMAP diet plus traditional dietary advice versus a low-carbohydrate diet versus pharmacological treatment in irritable bowel syndrome (CARIBS): a single-centre, single-blind, randomised controlled trial. Lancet Gastroenterol Hepatol. 2024 Jun;9(6):507-520. doi: 10.1016/S2468-1253(24)00045-1. Epub 2024 Apr 18. PMID 38643782
- [Derived] Nybacka S, Tornblom H, Simren M, Storsrud S. The Role of Carbohydrates in Irritable Bowel Syndrome: Protocol for a Randomized Controlled Trial Comparing Three Different Treatment Options. JMIR Res Protoc. 2022 Jan 17;11(1):e31413. doi: 10.2196/31413. PMID 35037893
- [Derived] Algera JP, Storsrud S, Lindstrom A, Simren M, Tornblom H. Gluten and fructan intake and their associations with gastrointestinal symptoms in irritable bowel syndrome: A food diary study. Clin Nutr. 2021 Oct;40(10):5365-5372. doi: 10.1016/j.clnu.2021.09.002. Epub 2021 Sep 9. PMID 34560607